CLINICAL TRIAL: NCT02040870
Title: A Phase I/II, Multicenter, Open-label, Single-arm Study of LDK378, Administered Orally in Adult Chinese Patients With ALK-rearranged (ALK-positive) Advanced Non-small Cell Lung Cancer (NSCLC) Previously Treated With Crizotinib Study Type: Interventional
Brief Title: LDK378 in Adult Chinese Patients With ALK-rearranged (ALK-positive) Advanced Non-small Cell Lung Cancer (NSCLC) Previously Treated With Crizotinib
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2109
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Results first posted 2019-01-17 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell lung Cancer; NSCLC; ALK; LDK378; ALK-rearranged; ALK-positive; advanced non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDK378 (Experimental): daily dosing, 28-day cycle patients
  Interventions: Drug: LDK378

INTERVENTIONS:
Drug: LDK378 — 750 mg once daily

SUMMARY:
A single-Arm, open-label, multi-center, phase I/II study in which the pharmacokinetics, safety, tolerability and efficacy of LDK378 will be assessed in adult Chinese patients with locally advanced or metastatic NSCLC harboring a confirmed ALK rearrangement. Patients must have demonstrated progression during or after crizotinib treatment whether or not previously treated with cytotoxic chemotherapy. Approximately 100 patients will be enrolled. For the first 15 patients enrolled in this study, patients will have an additional 5-day PK run-in period before treatment period. The pharmacokinetics profile of LDK378 in Chinese adult patients with ALK-rearranged NSCLC will be evaluated.

DETAILED DESCRIPTION:
This is a phase I/II, open-label, multi-center study in which the PK, safety, tolerability and efficacy of LDK378 will be assessed in adult Chinese patients with locally advanced or metastatic NSCLC harboring a confirmed ALK rearrangement (positive) as assessed using the Vysis ALK Break Apart FISH Probe Kit (Abbott Molecular Inc.) or positive as assessed by immunohistochemistry (IHC) test (Ventana Medical Systems, Inc) using rabbit monoclonal primary antibody assay (D5F3).

Patients must have demonstrated progression during or after crizotinib treatment whether or not previously treated with cytotoxic chemotherapy.

Approximately 100 patients with locally advanced or metastatic NSCLC which carry ALK -rearrangement will be enrolled in the study. The first 15 patients to be enrolled in the study will have PK sampling over 120-hour during the 5-day PK run-in period following a single oral dose at 750 mg. After the PK run-in period, the treatment period will start in which LDK378 will be given starting on Cycle 1 Day 1 in a continuous daily oral dosing in 28-day cycles. Separated from these 15 patients, the rest of the enrolled patients will receive LDK378 treatment at 750 mg QD on Cycle 1 Day 1.

Tumor response will be evaluated every 8 weeks (i.e. every 2 cycles) starting from the first day of treatment with LDK378 until the time of RECIST-defined PD by investigator assessment, withdrawal of consent for further follow-up, loss to follow-up or death.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC that carries an ALK rearrangement defined as positive using the FDA approved Vysis ALK Break Apart FISH Probe Kit (Abbott Molecular Inc.) test and scoring algorithm (including positivity criteria) or positive as assessed by the CFDA approved immunohistochemistry (IHC) test (Ventana Medical Systems, Inc)
* Age 18 years or older at the time of informed consent.
* Patients must have stage IIIB or IV NSCLC at the time of study entry and have had progressive disease during or after crizotinib treatment whether or not previously treated with cytotoxic chemotherapy. If treated with chemotherapy, maximum 2 lines are allowed.

Exclusion Criteria:

* Patients with known hypersensitivity to any of the excipients of LDK378
* Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms
* History of carcinomatous meningitis
* Presence or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years.
* clinically significant, uncontrolled heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-03-07 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- China (12):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guang Dong Province
  - Novartis Investigative Site, Guangzhou

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 100 patients were planned to be enrolled, and 103 patients were actually enrolled and analyzed.
Pre-assignment Details: Not Completed means that the participants discontinued from the treatment phase
Period: Overall Study
Arm/Group | LDK378
Started (Treatment Phase) | 103
Entered Post-treatment Follow-up | 2
Entered Survival Follow-up | 75
Discontinue From Study | 26
Completed | 0
Not Completed | 103
Not completed — Completed treatment phase | 6
Not completed — Adverse Event | 7
Not completed — Progressive disease | 58
Not completed — Physician Decision | 6
Not completed — Subject/guardian decision | 10
Not completed — Lost to Follow-up | 3
Not completed — Death | 13

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Arm/Group | LDK378
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
  Years | 49.3 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
  Participants
    Female | 48
    Male | 55
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
  Participants
    Chinese | 103

OUTCOME MEASURES:

1. Primary Outcome: Primary Pharmacokinetics (PK) Parameters of of LDK378 After Daily Oral Dose: AUClast, AUC0-24h, AUCinf
Description: AUClast: The area under the concentration-time curve from time zero to the last measurable concentration time.
  AUC0-24h: The area under the plasma concentration-time curve calculated from time zero to 24 hours.
  AUCinf: Area under the plasma (serum, or blood) concentration versus time curve from time zero to infinity
Time Frame: PK run-in phase (0h, 1h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 96h after PK run-in dose and predose Cycle 1 day 1 (C1D1)(approximately 120h after PK run in dose))
Population: The Pharmacokinetic Analysis Set (PAS) consists of all patients who receive at least one dose of LDK378 and provide at least one evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | LDK378
Number analyzed (Participants) | 103
ng*hr/mL
  AUClast: number analyzed (Participants) | 16
  AUClast | 10100 (52.6)
  AUC0-24h: number analyzed (Participants) | 16
  AUC0-24h | 3940 (49.6)
  AUCinf: number analyzed (Participants) | 14
  AUCinf | 11100 (57.7)

2. Primary Outcome: Primary Pharmacokinetics (PK) Parameter of of LDK378 After Daily Oral Dose: AUC0-24h
Description: AUC0-24h: The area under the plasma concentration-time curve calculated from time zero to 24 hours.
Time Frame: Cycle 2 Day 1 (after one cycle (28 days) of continous dosing)(0h, 1h, 2h, 3h, 4h , 6h , 8h and 24h)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | LDK378
Number analyzed (Participants) | 103
ng*hr/mL | 22000 (79.7)

3. Primary Outcome: Primary Pharmacokinetics (PK) Parameter of LDK378 After Daily Oral Dose: Cmax
Description: Cmax is the maximum (peak) concentration of drug in plasma
Time Frame: PK run-in phase (0h, 1h, 2h, 3h, 4h, 6h, 8h, 24h, 48h, 72h, 96h after PK run-in dose and predose Cycle 1 day 1 (C1D1)(approximately 120h after PK run in dose)) and C2D1(after one cycle (28 days) of continous dosing)(0h, 1h, 2h, 3h, 4h , 6h , 8h and 24h)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LDK378
Number analyzed (Participants) | 103
ng/mL
  PK run-in phase: number analyzed (Participants) | 16
  PK run-in phase | 233 (52.2)
  C2D1: number analyzed (Participants) | 14
  C2D1 | 1080 (78.0)

4. Primary Outcome: Primary Pharmacokinetics (PK) Parameter of LDK378 After Daily Oral Dose: Tmax
Description: Tmax is the time to reach maximum plasma concentration.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | LDK378
Number analyzed (Participants) | 103
hour
  PK run-in phase: number analyzed (Participants) | 16
  PK run-in phase | 5.94 [2.95 to 8.08]
  C2D1: number analyzed (Participants) | 14
  C2D1 | 5.88 [1.75 to 23.4]

5. Primary Outcome: Overall Summary of Adverse Events (AEs) - Per Occurence
Description: Safety and tolerability of LDK378 at 750 mg once daily dose in Chinese adult patients with ALK-rearranged locally advanced or metastatic NSCLC
Time Frame: up to 41 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Number; unit: occurrences
Arm/Group | LDK378
Number analyzed (Participants) | 103
occurrences
  All deaths | 65
  On-treatment deaths | 23
  Adverse Events (AEs) | 103
  AEs suspected to be drug related | 100
  Serious Adverse Events (SAEs) | 36
  SAEs suspected to be drug related | 7
  AEs leading to discontinuation | 15
  AEs requiring dose interruption | 34
  AEs requiring dose adjustment | 49
  AEs requiring dose adjustment or interruption | 64
  AEs requiring additional therapy | 94

6. Secondary Outcome: Overall Response Rate (ORR) Per RECIST 1.1 Per Investigator Assessment
Description: ORR calculated as the percentage of participants with a best overall response defined as complete response (CR) or partial response (PR). CR is the disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR is at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Number; unit: Percentage of participants
Arm/Group | LDK378
Number analyzed (Participants) | 103
Percentage of participants | 41.7

7. Secondary Outcome: ORR Per RECIST 1.1 Per Blind Independent Review Committee (BIRC) Assessment
Description: ORR per RECIST 1.1 calculated as the percentage of participants with a best overall response defined as complete response (CR) or partial response (PR). CR is the disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR is at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378
Number analyzed (Participants) | 103
Percentage of participants | 32.0 [23.2 to 42.0]

8. Secondary Outcome: Duration of Response (DOR) Per Investigator Assessment
Description: DOR, calculated as the time from the date of the first documented CR or PR to the first documented progression or all cause death. CR is the disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR is at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LDK378
Number analyzed (Participants) | 43
months | 7.5 [5.7 to 9.4]

9. Secondary Outcome: Disease Control Rate (DCR) Per Investigator Assessment
Description: DCR, calculated as the percentage of participants with best overall response of CR, PR, stable disease (SD) and Non-CR/Non-progressive disease (PD). CR is the disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR is at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. PD is at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition, the sum must also demonstrate an absolute increase of at least 5 mm. SD is neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD. Non-CR/Non-PD refers to best overall responses that are neither CR nor PD per RECIST 1.1 criteria for patients with non-measurable disease only at baseline.
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378
Number analyzed (Participants) | 103
Percentage of participants | 77.7 [68.4 to 85.3]

10. Secondary Outcome: Time to Response (TTR) Per Investigator Assessment
Description: TTR, calculated as the time from first dose of LDK378 to first documented response (CR+PR). CR is the disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR is at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Median (Full Range); unit: Months
Arm/Group | LDK378
Number analyzed (Participants) | 43
Months | 1.90 [1.6 to 12.9]

11. Secondary Outcome: Overall Intracranial Response Rate (OIRR) Per Investigator Assessment
Description: OIRR calculated as the ORR (CR+PR) of lesions in the brain for patients who have measureable disease in the brain at baseline. CR is the disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR is at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378
Number analyzed (Participants) | 23
Percentage of participants | 39.1 [19.7 to 61.5]

12. Secondary Outcome: Overall Intracranial Response Rate (OIRR) Per BIRC Assessment
Description: as for outcome 11
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378
Number analyzed (Participants) | 9
Percentage of participants | 0 [0.0 to 33.6]

13. Secondary Outcome: Progression Free Survival (PFS) Per Investigator Assessment
Description: PFS, defined as time from first dose of LDK378 to progression or death due to any cause.
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378
Number analyzed (Participants) | 103
Months | 7.2 [4.1 to 7.5]

14. Secondary Outcome: Overall Survival (OS)
Description: OS, defined as time from first dose of LDK378 to death due to any cause.
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378
Number analyzed (Participants) | 103
Months | 17.5 [10.8 to 24.3]

15. Secondary Outcome: Duration of Response (DOR) Per BIRC Assessment
Description: as for outcome 8
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LDK378
Number analyzed (Participants) | 33
months | 9.2 [7.3 to 14.7]

16. Secondary Outcome: Disease Control Rate (DCR) Per BIRC Assessment
Description: as for outcome 9
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378
Number analyzed (Participants) | 103
Percentage of participants | 67.0 [57.0 to 75.9]

17. Secondary Outcome: Time to Response (TTR) Per BIRC Assessment
Description: as for outcome 10
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Median (Full Range); unit: Months
Arm/Group | LDK378
Number analyzed (Participants) | 33
Months | 1.80 [1.6 to 3.7]

18. Secondary Outcome: Progression Free Survival (PFS) Per BIRC Assessment
Description: PFS, defined as time from first dose of LDK378 to progression or death due to any cause.
Time Frame: 40 months
Population: The Full Analysis Set (FAS) consisted of enrolled patients who received at least one dose of ceritinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378
Number analyzed (Participants) | 103
Months | 3.8 [3.6 to 5.6]

ADVERSE EVENTS:
Time Frame: Adverse Events are collected and reported from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to 41 months.
Arm/Group | LDK378
All-Cause Mortality (participants affected / at risk) | 23/103
Serious Adverse Events (participants affected / at risk) | 36/103
Other Adverse Events (participants affected / at risk) | 101/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDK378 (N=103)
Cardiac failure (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Impaired healing (General disorders) | 1
Lung infection (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Pulmonary mycosis (Infections and infestations) | 2
Post procedural oedema (Injury, poisoning and procedural complications) | 1
Blood bilirubin increased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureteric cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.0001% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDK378 (N=103)
Anaemia (Blood and lymphatic system disorders) | 36
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Angina pectoris (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Diplopia (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 10
Abdominal distension (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 22
Abdominal pain lower (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 30
Chronic gastritis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 77
Dry mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 4
Faecaloma (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 60
Oesophageal pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 63
Asthenia (General disorders) | 13
Chest discomfort (General disorders) | 4
Fatigue (General disorders) | 15
Gait disturbance (General disorders) | 1
Influenza like illness (General disorders) | 1
Malaise (General disorders) | 5
Non-cardiac chest pain (General disorders) | 22
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 1
Peripheral swelling (General disorders) | 2
Pyrexia (General disorders) | 20
Cholelithiasis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Gallbladder enlargement (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 2
Contrast media allergy (Immune system disorders) | 1
Abdominal infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 7
Respiratory tract infection (Infections and infestations) | 1
Tinea cruris (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 4
Ligament sprain (Injury, poisoning and procedural complications) | 1
Post procedural oedema (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 61
Amylase increased (Investigations) | 6
Apolipoprotein A-I decreased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 60
Bilirubin conjugated increased (Investigations) | 2
Blood albumin decreased (Investigations) | 11
Blood alkaline phosphatase (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 20
Blood bilirubin increased (Investigations) | 11
Blood calcium decreased (Investigations) | 1
Blood calcium increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 34
Blood glucose decreased (Investigations) | 1
Blood glucose increased (Investigations) | 9
Blood phosphorus decreased (Investigations) | 4
Blood potassium decreased (Investigations) | 4
Blood pressure increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Blood urea increased (Investigations) | 3
Blood uric acid increased (Investigations) | 2
Coagulation time prolonged (Investigations) | 1
Creatinine renal clearance decreased (Investigations) | 23
Creatinine renal clearance increased (Investigations) | 2
Electrocardiogram QT interval (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 9
Electrocardiogram T wave abnormal (Investigations) | 1
Electrocardiogram T wave inversion (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 27
Haemoglobin decreased (Investigations) | 9
Heart rate decreased (Investigations) | 1
Lipase increased (Investigations) | 2
Low density lipoprotein increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Lymphocyte percentage decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 7
Neutrophil count increased (Investigations) | 3
Neutrophil percentage increased (Investigations) | 2
Platelet count decreased (Investigations) | 11
Platelet count increased (Investigations) | 1
Prothrombin time prolonged (Investigations) | 1
Red blood cell count decreased (Investigations) | 2
Transaminases increased (Investigations) | 1
Weight decreased (Investigations) | 39
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 22
White blood cell count increased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 32
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 11
Hyponatraemia (Metabolism and nutrition disorders) | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureteric cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain oedema (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 12
Head discomfort (Nervous system disorders) | 1
Headache (Nervous system disorders) | 12
Hypoaesthesia (Nervous system disorders) | 3
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Eating disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 7
Chromaturia (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 5
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT02040870/SAP_000.pdf
  • Study Protocol (2015-10-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT02040870/Prot_001.pdf